CLINICAL TRIAL: NCT05931705
Title: Vit D Receptor Gene Polymorphism and Its Possible Association With Prevalence of Dental Caries
Brief Title: Vit D Receptor Gene Polymorphism
Acronym: VITAMIN D GENE
Status: Completed | Type: Observational
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, sudhir rama varma, Clinical Assistant Professor, Ajman University
Other Study IDs: (NU/CEC/2020/0339).
Record Dates: First submitted 2023-06-14; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Vitamin D Status
Keywords: Vitamin D Gene Polymorphism; Dental Caries; Cathelicidins
MeSH Terms: conditions — Dental Caries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High risk
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — questionnaire

SUMMARY:
The present cross-sectional observational study was conducted after the university ethical committee approved the research (NU/CEC/2020/0339). This study included 376 adults in the age group of 18-40Yrs. The patient information sheet briefed the study details and usage of salivary samples. Informed consent was obtained from participants. Healthy individuals free of associated systemic conditions, individuals not under any nutritional supplementation were included in the study, and lactating mothers, smokers, and menopausal women were excluded

DETAILED DESCRIPTION:
The present cross-sectional observational study was conducted after the university ethical committee approved the research (NU/CEC/2020/0339). This study included 376 adults in the age group of 18-40Yrs. The patient information sheet briefed the study details and usage of salivary samples. Informed consent was obtained from participants. Healthy individuals free of associated systemic conditions, individuals not under any nutritional supplementation were included in the study, and lactating mothers, smokers, and menopausal women were excluded.

Further, the subjects were divided into active and caries-free based on caries experience. Two indexing methods were utilized to record the decay status, i.e., Decay, Missing, filled (DMFT) and Pulpal, Ulcerative, Fistula (PUFA) scores. Caries active group was further divided into a High-risk group (DMFT=< 10), Moderate risk (DMFT= 4-9), and Low risk (DMFT=1-3).

Questionnaire: Baseline information was gathered, including specifics on age, sex, height, weight, dietary preferences (non-veg/veg), and dental hygiene practices.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals free of associated systemic conditions
* Individuals not under any nutritional supplementation

Exclusion Criteria:

* lactating mothers
* smokers
* menopausal women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population included participants with active dental caries and associated wasting disease of the teeth due to caries
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
DMFT scores | six months
  Scores are 1 for dental caries present and 0 for dental caries absent

CONTACTS AND LOCATIONS:
Locations (1):
- AB shetty Institute of dental sciences, Mangaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
Results
Supporting Information: Study Protocol, SAP, ICF, CSR